CLINICAL TRIAL: NCT01758627
Title: The Role of Peritoneal Dialysis in Patients With Refractory Heart Failure and Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2012-0750
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2016-04

CONDITIONS: Refractory Heart Failure; Chronic Kidney Disease
Keywords: Peritoneal dialysis,; chronic kidney disease,; refractory heart failure
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic | interventions — Peritoneal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peritoneal dialysis group (No Intervention)
- Conventional treatment group (Experimental): medical treatment such as diuretics
  Interventions: Drug: Peritoneal dialysis (PD)

INTERVENTIONS:
Drug: Peritoneal dialysis (PD) — PD exchanges will be customized depending on patient fluid status. At least one daily exchange of icodextrin PD solution will be provided to PD group.
  Other Names: PD exchanges will be customized depending on patient fluid status. At least one daily exchange of icodextrin PD solution will be provided to PD group.
  Arms: Conventional treatment group

SUMMARY:
In patients with advanced heart failure (HF), systemic congestion is the main indication for hospitalization. Recent evidence has highlighted the role of fluid retention in the pathogenesis of renal dysfunction and subsequent diuretic resistance. Previous kidney disease, diuretic resistance, and progression of renal dysfunction often coexist in patients with HF and persistent volume overload. This clinical presentation represents the most extreme feature of the cardio-renal syndrome. However, available therapeutic options for this ominous condition are scarce and limited. Indeed, there are no data from randomized control trials using pharmacological interventions that support the beneficial effect on survival. Interestingly, intermittent ultrafiltration has recently emerged as an alternative therapeutic option for reducing volume overload in patients with refractory HF. Current literature suggests that it has potential advantages over standard medical treatment particularly in acute stages of HF. Among ultrafiltration methods, peritoneal dialysis (PD) has been preferred as an additional resource for the treatment of advanced congestive heart failure (CHF) compared with hemodialysis because it can provide a more physiological and continuous ultrafiltration. In fact, several studies showed that use of PD improved clinical functional class and hemodynamic parameters and reduced hospitalization rates in patients with CHF. Nevertheless, most studies were limited by retrospective analyses of small sample size, prospective observational design with no control group, or inclusion of patients with end-stage renal failure. Therefore, well-designed prospective randomized controlled studies are mandatory to confirm the effects of PD in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. At least two non-planned admissions for acute heart failure (AHF), the last episode being in the past 6 months
2. New York Heart Association (NYHA) functional class III/IV and left ventricular ejection fraction (LVEF) less than 40%
3. Persistent congestion despite optimal loop diuretic therapy
4. Presence of renal dysfunction [estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2] documented at least once in the last 6 months

Exclusion Criteria:

1. < 20 years of age
2. Pregnancy
3. Unsuitable for PD (patients with major abdominal wall defects)
4. Allergic to starch or other contraindication to icodextrin (5) End-stage renal disease (eGFR < 10 ml/min/1.73 m2) requring dialysis treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10-08 (Actual); Study Completion 2015-10-08 (Actual)

PRIMARY OUTCOMES:
Changes of New York Heart Association (NYHA) functional class | at 0 (±1 week), 12 (±1 week), and 24 (±1 week) weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Nephrology, Department of Internal Medicine Yonsei University College of Medicine, Seoul, South Korea